CLINICAL TRIAL: NCT04355247
Title: Prophylactic Corticosteroid to Prevent COVID-19 Cytokine Storm
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Auxilio Mutuo Cancer Center (Other)
Responsible Party: Principal Investigator, Fernando Cabanillas, Medicine Doctor/Medical Director, Auxilio Mutuo Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CCAM 20-01
Record Dates: First submitted 2020-04-17; First posted 2020-04-21 (Actual); Last update posted 2020-04-21 (Actual); Status verified 2020-04

CONDITIONS: Covid-19
Keywords: Severe Acute Respiratory Syndrome (SARS)-Cov-2 Virus
MeSH Terms: conditions — COVID-19; Severe Acute Respiratory Syndrome | interventions — Methylprednisolone

STUDY DESIGN:
Intervention Model Description: This is a pilot Phase II exploratory study. It is a non-randomized study which will be carried out at Auxilio Mutuo Hospital and possibly at other institutions to be recruited.
  The investigator plans to enter a total of 20 patients in order to determine whether the risk of progressing to respiratory failure can be reduced by administering corticosteroids.
  The investigator assume that virtually all patients who met the criteria for entry into this trial will develop respiratory insufficiency if left untreated.
  If </= 50% of patients with high risk develop respiratory failure the investigator will consider the treatment as successful.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm (Experimental): * Patients will be admitted to a regular room in the hospital (not ICU)
  * They will be monitored closely with vital signs every 4 hours to ensure their respiratory and cardiovascular status do not deteriorate.
  * Methylprednisolone 80 mg IV bolus injection will be given daily x 5 days starting upon day 1 of admission to hospital.
  Interventions: Drug: MethylPREDNISolone 80 Mg/mL Injectable Suspension

INTERVENTIONS:
Drug: MethylPREDNISolone 80 Mg/mL Injectable Suspension — * Patients will be admitted to a regular room in the hospital (not ICU)
  * They will be monitored closely with vital signs every 4 hours to ensure their respiratory and cardiovascular status do not deteriorate.
  * Methylprednisolone 80 mg IV bolus injection will be given daily x 5 days starting upon day 1 of admission to hospital.

SUMMARY:
This is a Phase II pilot exploratory study designed to investigate if prophylactic treatment with short term steroids administered to high risk Covid-19 patient might prevent cytokine storm and progression to respiratory failure. High risk is defined based on serologic markers of inflammation that include abnormalities of Interleukin 6 (IL-6), Ferritin , D-dimer, Lactate Dehydrogenase (LDH), as well as lymphopenia and impaired O2 saturation prior to or on the 7th day of first symptom of Covid-19.

DETAILED DESCRIPTION:
To decrease the rate of progression to hypoxemic respiratory failure in high risk patients with Covid-19, treated with prophylactic steroids during the first phase of the disease.

ELIGIBILITY:
Inclusion Criteria:

* All patients diagnosed with Covid-19 will be registered on the study regardless pf their severity, but only those who meet high risk criteria will be treated with steroids. Those who don't meet the criteria will only be registered with no need to collect further data except baseline labs and CT Chest. They should sign the consent form and the data manager can collect the rest of the information.
* Patients older than 18 years diagnosed with Covid-19 by Polymerase Chain Reaction (PCR) or by rapid serological test will be eligible. Cases who are Immunoglobulin G (IgG) positive but Immunoglobulin M (IgM) negative, will not be considered eligible unless they are positive for molecular PCR test. Eligible patients will be registered on study on or before 7 days from first onset of symptoms.

Exclusion Criteria:

* Any patient with life expectancy < 1 month
* Any patient who is oxygen dependent
* Any patient with long standing history of severe Chronic Obstructive Pulmonary Disease (COPD)
* Any patient who is chronically oxygen dependent because of previous existing lung disease
* Anyone with severely uncontrolled diabetes despite adequate management
* Anyone with active serious bacterial infection such as septicemia or pneumonia
* Anyone receiving Tocilizumab (anti IL-6 therapy) or plasma therapy
* Any patient already receiving steroids from another pre-existing illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-04-14 (Actual); Primary Completion 2020-07-31 (Estimated); Study Completion 2021-04-30 (Estimated)

PRIMARY OUTCOMES:
Clinical complete response criteria | 14 days
  Clinical complete response criteria requires all the following:
  * No need for ventilatory support at any point
  * O2 Saturation of >/= 93% by day 14 of therapy
  * Alive by day 28 from registration
  * CT chest with minimal or no evidence of disease by day 28 from registration
Clinical Partial Response criteria | 14 days
  Clinical Partial Response criteria require that 2 of the following be present by day 14 of therapy:
  * No need for ventilatory support at any point O2 saturation > 93% bay day 14 from registration
  * CT chest stable to improve over baseline by day 28 from registration

SECONDARY OUTCOMES:
Secondary response criteria | 14 days
  Decrease of at least 25% in anyone of the following markers: IL-6, Ferritin, D-dimer, C reactive protein (CRP) or LDH by day 14
  - Improvement of absolute lymphocyte count in those presenting with lymphopenia. Improvement is defined as increase by 25% or more by day 14.

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Cabanillas, MD, Principal Investigator — Hospital Español Auxilio Mutuo
Locations (2):
- Puerto Rico (2):
  - Hospital Auxilio Mutuo Cancer Center, San Juan, PR
  - San Juan City Hospital / Puerto Rico Medical Center, San Juan

REFERENCES:
- [Background] Gautret P, Lagier JC, Parola P, Hoang VT, Meddeb L, Mailhe M, Doudier B, Courjon J, Giordanengo V, Vieira VE, Tissot Dupont H, Honore S, Colson P, Chabriere E, La Scola B, Rolain JM, Brouqui P, Raoult D. RETRACTED: Hydroxychloroquine and azithromycin as a treatment of COVID-19: results of an open-label non-randomized clinical trial. Int J Antimicrob Agents. 2020 Jul;56(1):105949. doi: 10.1016/j.ijantimicag.2020.105949. Epub 2020 Mar 20. PMID 32205204
- [Background] Chen L, Xiong J, Bao L, Shi Y. Convalescent plasma as a potential therapy for COVID-19. Lancet Infect Dis. 2020 Apr;20(4):398-400. doi: 10.1016/S1473-3099(20)30141-9. Epub 2020 Feb 27. No abstract available. PMID 32113510
- [Background] Carr AC. A new clinical trial to test high-dose vitamin C in patients with COVID-19. Crit Care. 2020 Apr 7;24(1):133. doi: 10.1186/s13054-020-02851-4. No abstract available. PMID 32264963
- [Background] Zhou F, Yu T, Du R, Fan G, Liu Y, Liu Z, Xiang J, Wang Y, Song B, Gu X, Guan L, Wei Y, Li H, Wu X, Xu J, Tu S, Zhang Y, Chen H, Cao B. Clinical course and risk factors for mortality of adult inpatients with COVID-19 in Wuhan, China: a retrospective cohort study. Lancet. 2020 Mar 28;395(10229):1054-1062. doi: 10.1016/S0140-6736(20)30566-3. Epub 2020 Mar 11. PMID 32171076
- [Background] Zhang C, Wu Z, Li JW, Zhao H, Wang GQ. Cytokine release syndrome in severe COVID-19: interleukin-6 receptor antagonist tocilizumab may be the key to reduce mortality. Int J Antimicrob Agents. 2020 May;55(5):105954. doi: 10.1016/j.ijantimicag.2020.105954. Epub 2020 Mar 29. PMID 32234467
- [Background] Wu C, Chen X, Cai Y, Xia J, Zhou X, Xu S, Huang H, Zhang L, Zhou X, Du C, Zhang Y, Song J, Wang S, Chao Y, Yang Z, Xu J, Zhou X, Chen D, Xiong W, Xu L, Zhou F, Jiang J, Bai C, Zheng J, Song Y. Risk Factors Associated With Acute Respiratory Distress Syndrome and Death in Patients With Coronavirus Disease 2019 Pneumonia in Wuhan, China. JAMA Intern Med. 2020 Jul 1;180(7):934-943. doi: 10.1001/jamainternmed.2020.0994. PMID 32167524
- [Background] Russell CD, Millar JE, Baillie JK. Clinical evidence does not support corticosteroid treatment for 2019-nCoV lung injury. Lancet. 2020 Feb 15;395(10223):473-475. doi: 10.1016/S0140-6736(20)30317-2. Epub 2020 Feb 7. No abstract available. PMID 32043983
- [Background] Grein J, Ohmagari N, Shin D, Diaz G, Asperges E, Castagna A, Feldt T, Green G, Green ML, Lescure FX, Nicastri E, Oda R, Yo K, Quiros-Roldan E, Studemeister A, Redinski J, Ahmed S, Bernett J, Chelliah D, Chen D, Chihara S, Cohen SH, Cunningham J, D'Arminio Monforte A, Ismail S, Kato H, Lapadula G, L'Her E, Maeno T, Majumder S, Massari M, Mora-Rillo M, Mutoh Y, Nguyen D, Verweij E, Zoufaly A, Osinusi AO, DeZure A, Zhao Y, Zhong L, Chokkalingam A, Elboudwarej E, Telep L, Timbs L, Henne I, Sellers S, Cao H, Tan SK, Winterbourne L, Desai P, Mera R, Gaggar A, Myers RP, Brainard DM, Childs R, Flanigan T. Compassionate Use of Remdesivir for Patients with Severe Covid-19. N Engl J Med. 2020 Jun 11;382(24):2327-2336. doi: 10.1056/NEJMoa2007016. Epub 2020 Apr 10. PMID 32275812
- See also: The potential role of IL-6 in monitoring severe case of coronavirus disease 2019 — https://www.medrxiv.org/content/10.1101/2020.03.01.20029769v2
- See also: Level of IL-6 predicts respiratory failure in hospitalized symptomatic COVID-19 patients — https://www.medrxiv.org/content/10.1101/2020.04.01.20047381v2